CLINICAL TRIAL: NCT01367288
Title: Comparative Study of Neoadjuvant Chemotherapy With and Without Zometa for Management of Locally Advanced Breast Cancers
Acronym: NEOZOL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009.568
Record Dates: First submitted 2010-09-17; First posted 2011-06-07 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2014-05

CONDITIONS: Locally Advanced Breast Cancer; Ductal Histologic Type; Without Her 2 Overexpression
Keywords: locally advanced breast cancer; neoadjuvant chemotherapy; HER2-negative breast cancer; stage IIb breast cancer; stage IIIa breast cancer; Zoledronic acid; bisphosphonate; zometa; therapeutic response; VEGF serum; tumors markers; neoangiogenesis; apoptosis; proliferation; disseminated tumors cells; gamma-delta T cells activation
MeSH Terms: conditions — Breast Neoplasms; Neovascularization, Pathologic | interventions — Zoledronic Acid; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Neoadjuvant therapy + Zometa) (Experimental): Patients will be treated every 3 weeks (+/- 2 days ) for 8 cycles in total. The 4 first cycles : Zometa 4 mg (in a 15 min. infusion) + doxorubicin (60 mg/m²) + cyclophosphamide (600 mg/m²). The 4 last cycles with Zometa 4 mg (in a 15 min. infusion) + docetaxel (100 mg/m²)
  Interventions: Drug: Zometa + Neoadjuvant therapy; Drug: Neoadjuvant therapy
- B (Neoadjuvant therapy) (Active Comparator): Patients will be treated every 3 weeks (+/- 2 days) for 8 cycles in total. The 4 first cycles : doxorubicin (60 mg/m²) combined with cyclophosphamide (600 mg/m²). The 4 last cycles with docetaxel (100 mg/m²)
  Interventions: Drug: Neoadjuvant therapy

INTERVENTIONS:
Drug: Zometa + Neoadjuvant therapy — 4 mg (in a 15 min. infusion) every 3 weeks for a total of 8 injections
  Arms: A (Neoadjuvant therapy + Zometa)
Drug: Neoadjuvant therapy — 4 injections of doxorubicin (60 mg/m²) combined with cyclophosphamide (600 mg/m²) every 3 weeks (+/- 2 days), followed by 4 injections of docetaxel (100 mg/m²) every 3 weeks (+/- 2 days)

SUMMARY:
Breast cancer is the leading female cancer by a very wide margin in France. Despite widespread breast cancer screening, many cases of breast cancer are discovered at a locally advanced stage. The tumoral consequences of a cancer size greater than 3 cm are: increased risk of metastasis and death and, most often, impossibility of performing breast-conserving surgery (a mastectomy is usually advisable in case of a first surgical procedure). It is increasingly recommended to treat locally advanced breast cancers with neoadjuvant chemotherapy. Very numerous studies have shown that by proceeding that way, the oncologic prognosis was not harmed and, on the contrary, it was possible to obtain sufficient tumor response to allow breast-conserving treatment in more than 60% of cases.

The use of zoledronic acid (Zometa) has an established place in the management of malignancies with a predilection for skeletal involvement (in particular metastasis). Although the main target of biphosphonates is the osteoclast, there is also preclinical data indicating that biphosphonates can have effects on cells other than osteoclasts, including tumor cells. Anti-tumor activity including inhibition of tumor cell growth and induction of tumor cell apoptosis, inhibition of tumor cell adhesion and invasion, and anti-angiogenic effects have been demonstrated. In addition several in vitro studies have shown that Zometa causes synergistic induction of breast cancer cell apoptosis when combined with clinically relevant concentrations of chemotherapy drugs such as paclitaxel and doxorubicin. Therefore testing of combinations of biphosphonates with these agents in breast cancer is of significant interest.

In the context of locally advanced breast cancers, the combination of a bisphosphonate with neoadjuvant chemotherapy appears to have an important potential: preventing possible bone metastases, but also possibly amplifying the efficacy of the chemotherapy's tumoricidal activity, both on the primary tumor and on potential metastatic localizations.

So it appears that, the use of bisphosphonates in a neoadjuvant situation presents a potentially favorable benefit-risk ratio. That is why we are proposing to perform a prospective randomized multicenter comparative study to evaluate 2 systemic neoadjuvant treatments, one with Zometa and the other without Zometa, in patients with locally advanced breast cancer. Zometa will be administered according to the usual administration procedure: one infusion every 3 weeks.

The therapeutic response will be evaluated by studying the different biological markers (circulating blood and bone marrow tumor cells, serum cell apoptosis and neoangiogenesis markers, bone resorption markers, etc.), but also by analyzing clinical, radiologic, and histologic response and by breast conservation rates. The impact of other factors that may affect therapeutic response will be taken into account: aggressivity of the tumor, presence or absence of tumor receptors, tumor stage, etc.

The purpose of the study is to show a marked benefit of treatment with Zometa in managing locally advanced breast cancers with synergistic action of the neoadjuvant chemotherapy and improvement in the laboratory parameters of tumor aggressivity. These markers will be used as surrogate markers of long term outcome.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older
* Absence of contraindication to treatment with Zometa: creatinine clearance greater than 30 mL/min (with Cockroft or MDRD method).
* Breast cancer (TNM IIa, IIb, IIIa) larger than 2cm in maximal diameter able to benefit from neoadjuvant chemotherapy
* Ductal or lobular histological type of the breast tumor
* WHO performance status 0-2
* Patient who understands the french language
* Covered by, or having the right to Social Security
* Signed informed consent

Exclusion Criteria:

* Breast cancers of rare histological type (other than ductal and lobular)
* Noninvasive cancer
* Multifocal tumor (more than 2 tumoral lesions or 2 tumoral lesions distant more than 2cm each other)
* T4 breast tumor
* Presence of organ, bone, or skin metastases (in the initial staging workup)
* Patient with a history of breast cancer
* Other cancer currently in treatment (except carcinoma in situ).
* Severe systemic disease potentially interfering with follow-up.
* Contraindication to injected products: known allergy to bisphosphonates, zoledronic acid or excipients, severe renal failure (creatinine clearance < 30 mL/min with Cockroft or MDRD method).
* Women who are pregnant (positive pregnancy test) or breast-feeding, or absence of contraception in a woman who is able to become pregnant.
* Patient with evolutionary dental problems, including dental infection or infection of the jaw,intrabuccal exposure of jawbone, and history or current diagnosis of osteonecrosis of the jaw,requiring a fast chirurgical care.
* Prior treatment with bisphosphonates (either IV or oral).
* History of severe bone disease (severe osteoporosis with multiple skeletal-related events).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Decrease in serum VEGF concentration treatment | 8 months
  To assess the improvement obtained by adding Zometa treatment to neoadjuvant chemotherapy in patients with locally advanced breast cancer on concentrations of serum VEGF (neoangiogenesis marker and prognostic factor) before treatment and during surgery after neoadjuvant treatment (i.e., at about 8 months)

SECONDARY OUTCOMES:
Change in CTC | 8 months
  To assess the impact of each of the treatment arms on circulating tumor cells (CTC) present in the blood
Change in serum markers of apoptosis | every 3 weeks during 8 months
  To assess the impact of each of the treatment arms on serum markers of apoptosis,
Change in serum tumor markers | every 3 weeks during 8 monthes
  assessment of the change in serum tumor markers by CEA, V-EGF and CA 15-3 assay
Change in tumor markers of apoptosis and proliferation | before treatment, at 90-105 days and at surgical excision
Change in circulating gamma-delta T-cell activation | every 3 weeks during 8 monthes
Therapeutic complications | at each of the chemotherapy sessions and during the final surgery
  Assessment of renal failure and osteonecrosis of the jaw
Assessment of tumor response | at the start of treatment, at day 90-105, after 4 neoadjuvant treatment sessions, after all 8 neoadjuvant chemotherapy sessions
  To assess the impact of each of the strategies treatment arms on clinical, and radiological tumour response (maximum tumour diameter)
Assessment of histological tumor response | during the final surgery
Breast conservation rate | during the final surgery
  To assess the breast conservation rate for each of the strategies
Assessment of the intermediate tumor response | at day 90-105
  To assess the changes in tissue biomarkers at day 90-105 (intermediate biopsy) in each of the strategies.
Assessment of the markers studied in the complementary study | at the end of the treatment
  * measurement of IPP and ApppI (PBMCs), FPPS mRNA (PBMCs)
  * FACS analysis of gamma-delta T cell subsets, measurement of IFNg, TNFa
  * Measurement of gamma-delta T cells cytotoxic activity
  * Injection of expanded gamma-delta T cells in NOD/SCID mice bearing patients' tumors and follow-up of animals (tumor size measurement, survival, IHC). Correlation with clinicopathological factors and clinical outcome of patients.
  * RNA extraction of primary tumour biopsies before treatment and at the time of surgery for DNA microarray hybridization studies

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Mathevet, Professor, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hopital Femme Mère Enfant, Service de Gynécologie, Bron, France

REFERENCES:
- [Result] Lelievre L, Clezardin P, Magaud L, Roche L, Tubiana-Mathieu N, Tigaud JD, Topart D, Raban N, Mouret-Reynier MA, Mathevet P. Comparative Study of Neoadjuvant Chemotherapy With and Without Zometa for Management of Locally Advanced Breast Cancer With Serum VEGF as Primary Endpoint: The NEOZOL Study. Clin Breast Cancer. 2018 Dec;18(6):e1311-e1321. doi: 10.1016/j.clbc.2018.07.005. Epub 2018 Jul 10. PMID 30098917
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716